CLINICAL TRIAL: NCT03957278
Title: A Prospective, Multi-Center, Single Arm Study to Evaluate the DAISe System During Neurointervention for Acute Ischemic Stroke
Brief Title: A Study to Evaluate the DAISe System During Neurointervention for Acute Ischemic Stroke
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Device modifications
Sponsor: MIVI Neuroscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101361
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Stroke, Acute
Keywords: Mechanical thrombectomy; Acute ischemic stroke; neurovascular intervention
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Single arm, multi-center, prospective study where all eligible subjects are treated with the study device after enrollment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DAISe System (Experimental): The DAISe System consists of the DAISe thrombectomy device used in with the Q Aspiration Catheter.
  Interventions: Device: DAISe System

INTERVENTIONS:
Device: DAISe System — The DAISe System is indicated for revascularization of patients with acute ischemic stroke for the removal of fresh thrombi from vessels in the neurovasculature.

SUMMARY:
This purpose study is to demonstrate the safety and performance of the DAISe System used to remove clot in the brain during a stroke. This study will assess how well the device removes clot from the brain and how well patients recover from their stroke. This study plans to enroll 100 study patients at up to 10 hospitals in Europe. Study patients are followed for 3 months after the procedure.

DETAILED DESCRIPTION:
The study is a prospective, multi-center, single arm study that will enroll a maximum of 90 subjects, plus up to 50 roll-in subjects. A maximum of 10 sites in Europe will be involved in this study. The primary performance endpoint is successful revascularization defined as TICI 2b-3 flow in the target vessel post-treatment of up to three passes with the DAISe System. The primary safety endpoint is symptomatic intracranial haemorrhage at 24 hours post-procedure as detected by CT/MRI with an NIHSS change of >/=4. Subject will be followed through hospital discharge with a visit at Day 1 post procedure, Day 7 or prior to discharge/transfer, 30 days and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 85 years.
* Diagnosis of acute ischemic stroke with study enrollment time < 8 hours from onset of symptoms.
* Disabling stroke defined as a baseline NIHSS > 6.
* Pre-stroke (24 hours prior to stroke onset) independent functional status in activities of daily living with modified Rankin Score 0-1.
* If thrombolytic therapy (tPA) is administered, it must be administered per the prescribing information.
* Confirmed symptomatic intracranial occlusion, based on single phase, multiphase or dynamic CTA, at one or more of the following locations: Carotid T/L, M1 MCA, or M1-MCA equivalent (2 or more M2-MCAs), or M2-MCA.
* The following baseline imaging criteria should be met: MRI criterion: ASPECTS Score > 4 OR CT criterion: ASPECTS > 6
* Signed informed consent from patient or legally authorized representative.

Exclusion Criteria:

* CT or MRI evidence of recent/ fresh hemorrhage on presentation.
* Clinical history, past imaging or clinical judgment suggests that the intracranial occlusion is chronic.
* Rapidly improving neurological deficits based on the investigator's clinical judgement.
* Pregnancy
* Severe contrast allergy or absolute contraindication to iodinated contrast.
* No femoral pulses or very difficult endovascular access that will result in an inability to deliver endovascular therapy.
* Evidence of dissection in the carotid or middle cerebral arteries.
* Severe unilateral or bilateral carotid artery stenosis requiring treatment at the time of the procedure as determined during diagnostic angiography.
* Renal failure (serum creatinine level ≥ 4 mg/dL or on dialysis).
* Severe, sustained hypertension (SBP >185 mmHg or DBP >110 mmHg).
* Cerebral vasculitis.
* Suspicion of aortic dissection, presumed septic embolus or suspicion of bacterial endocarditis.
* Clinical symptoms suggestive of bilateral stroke or occlusions in multiple vascular territories (e.g., bilateral anterior circulation, or anterior/posterior circulation).
* Seizure due to stroke.
* Platelet count < 50,000/mm3.
* A severe or fatal comorbid illness that will prevent improvement or follow-up or that will render the procedure unlikely to benefit the patient.
* Patient is unable or unwilling complete follow up visits.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2021-11-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with successful revascularization | intra-procedural
  Defined as mTICI 2b-3 flow in the target vessel post-treatment of up to three passes with the DAISe System.
Rate of symptomatic intracranial haemorrhage | 12-36 hours post procedure
  24 hours post-procedure as detected by CT/MRI with an NIHSS change of >4

SECONDARY OUTCOMES:
Number of participants with successful revascularization of mTICI 2b-3 as a result of the first attempt with the DAISe System | intra-procedural
Number of participants with successful revascularization of mTICI 3 as a result of the first attempt with the DAISe System | intra-procedural
Number of participants with successful revascularization of final mTICI 2b-3 at the end of the procedure | intra-procedural
Time from groin puncture to successful revascularization defined as final mTICI 2b-3 flow | intra-procedural
Rate of procedure-related complications | post procedure through discharge
Rate of embolization to a new vascular territory (ENT) | intra-procedural
Good functional outcome for participants measured by Modified Rankin Scale score of 0-2. | 30 days and 3 months post procedure
  The Modified Rankin Scale (mRS) measures neurological disability or dependence for stroke patients on a scale of 0 (no symptoms) to 6 (deceased).
Quality of life for participants: PROMIS Scale | 3 months post procedure
  PROMIS Scale
Rate of all cause mortality | 30 days and 3 months post procedure

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Erasme Hospital, Brussels
  - Hospital Civil Marie Curie, Charleroi

IPD SHARING:
Plan to Share IPD: No